CLINICAL TRIAL: NCT04171388
Title: Enhancing Nutrition and Antenatal Infection Treatment for Maternal and Child Health in Amhara Region, Ethiopia
Brief Title: Enhancing Nutrition and Antenatal Infection Treatment for Maternal and Child Health in Ethiopia
Acronym: ENAT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Trial withdrawn due to COVID-19.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Addis Continental Institute of Public Health (Other); Johns Hopkins Bloomberg School of Public Health (Other); Boston Children's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Harvard School of Public Health (HSPH) (Other); Amhara Public Health Institute (Unknown); Jhpiego (Other)
Responsible Party: Principal Investigator, Anne Lee, Pediatric Hospitalist, Director of Global Newborn Health, Department of Pediatric Newborn Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018P002479
Record Dates: First submitted 2019-10-09; First posted 2019-11-20 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Low Birthweight; Preterm Birth; Maternal; Malnutrition, Affecting Fetus; Sexually Transmitted Diseases; Urinary Tract Infections; Pregnancy and Infectious Disease
Keywords: Low birthweight; Preterm birth; Maternal nutrition; Small for gestational age; Chlamydia; Gonorrhea; Urinary tract infection; Presumptive antibiotics
MeSH Terms: conditions — Premature Birth; Malnutrition; Sexually Transmitted Diseases; Urinary Tract Infections; Communicable Diseases; Chlamydia Infections; Gonorrhea | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: 2x3 factorial randomized controlled trial, with cluster randomization of nutrition interventions and individually randomized infection management interventions
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking of Azithro vs. Placebo arm only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Routine care: Placebo (Placebo Comparator): In all pregnancies presenting at all centers, routine antenatal care will be strengthened:
  * Provision of iron-folic acid and tetanus toxoid vaccine
  * Screening for anemia and blood pressure
  * Screening/treatment of HIV, syphilis, malaria, tuberculosis
  Placebo tablets will be administered twice in pregnancy: at enrollment (<=24 weeks) and a follow up ANC visit at least 4 weeks later.
  Interventions: Drug: Placebo oral tablet 500 mg
- Routine care: Azithromycin (Experimental): Azithromycin will be provided twice in pregnancy: at enrollment (<=24 weeks) and a follow up ANC visit at least 4 weeks later.
  Interventions: Drug: Azithromycin 500 mg
- Routine care: Enhanced Infection Management Package (EIMP) (Experimental): At the study enrollment visit, pregnant women will receive presumptive deworming (albendazole) and screening for urinary tract infection and sexually transmitted infections (chlamydia and gonorrhea). Women with identified infections will be treated with appropriate antibiotics. A second dose of albendazole will be given at a follow up ANC visit at least 4 weeks after enrollment.
  Interventions: Other: Enhanced Infection Management Package (EIMP)
- Enhanced Nutrition Package (ENP): Placebo (Experimental): Pregnant women will receive a daily multiple micronutrient. Women with undernutrition, identified with mid-upper arm circumference <23 cm, will receive a daily fortified balanced energy protein supplement.
  Placebo tablets will be administered twice in pregnancy: at enrollment (<=24 weeks) and a follow up ANC visit at least 4 weeks later.
  Interventions: Dietary Supplement: Multiple Micronutrient or Fortified Balanced Energy Protein Supplement; Drug: Placebo oral tablet 500 mg
- ENP: Azithromycin (Experimental): Pregnant women will receive a daily multiple micronutrient. Women with undernutrition, identified with mid-upper arm circumference <23 cm, will receive a daily fortified balanced energy protein supplement.
  Azithromycin will be provided twice in pregnancy: at enrollment (<=24 weeks) and a follow up ANC visit at least 4 weeks later.
  Interventions: Drug: Azithromycin 500 mg; Dietary Supplement: Multiple Micronutrient or Fortified Balanced Energy Protein Supplement
- ENP: EIMP (Experimental): Pregnant women will receive a daily multiple micronutrient. Women with undernutrition, identified with mid-upper arm circumference <23 cm, will receive a daily fortified balanced energy protein supplement.
  At the study enrollment visit, pregnant women will receive presumptive deworming (albendazole) and screening for urinary tract infection and sexually transmitted infections (chlamydia and gonorrohea). Women with identified infections will be treated with appropriate antibiotics. A second dose of albendazole will be given at a follow up ANC visit at least 4 weeks after enrollment.
  Interventions: Dietary Supplement: Multiple Micronutrient or Fortified Balanced Energy Protein Supplement; Other: Enhanced Infection Management Package (EIMP)

INTERVENTIONS:
Drug: Azithromycin 500 mg — Azithromycin 500mg (Kern Pharma): 2g (4 tablets) at 2 time points during pregnancy: enrollment (<=24 weeks gestation), and follow-up ANC at least 4 weeks later
  Arms: ENP: Azithromycin; Routine care: Azithromycin
Dietary Supplement: Multiple Micronutrient or Fortified Balanced Energy Protein Supplement — Daily multiple micronutrient (MMN) tablet (Contract Pharmacal Corp) for women with mid-upper arm circumference (MUAC) >=23 cm, OR Daily fortified balanced energy protein (BEP) supplement (DSM South Africa; Faffa Food Products): Fortified corn-soy blend (784 kcal/day) for women with MUAC <23 cm
  Arms: ENP: Azithromycin; ENP: EIMP; Enhanced Nutrition Package (ENP): Placebo
Drug: Placebo oral tablet 500 mg — Placebo 500mg (Idifarma): 2g (4 tablets) at 2 time points during pregnancy; enrollment (<24 weeks gestation), and follow up ANC at least 4 weeks later
  Arms: Enhanced Nutrition Package (ENP): Placebo; Routine care: Placebo
Other: Enhanced Infection Management Package (EIMP) — ENROLLMENT VISIT: Screening for bacteriuria with urine culture, and antimicrobial susceptibility testing; Screening for chlamydia and gonorrhea with Cepheid GeneXpert; Presumptive deworming with albendazole 500mg.
  FOLLOWUP TREATMENT VISIT: For women with identified urinary tract infection or asymptomatic bacteriuria, treatment with antibiotics based on antimicrobial susceptibility patterns. For women with identified chlamydia or gonorrhea, treatment of woman (and partner) with appropriate antibiotics. Test of cure sample and retreatment of infection.
  Second deworming with albendazole at least 4 weeks after enrollment ANC visit.
  Arms: ENP: EIMP; Routine care: Enhanced Infection Management Package (EIMP)

SUMMARY:
The ENAT study will test the impact of packages of antenatal interventions to enhance maternal nutrition and manage pregnancy infections on the outcomes of infant birth size, gestational length, and infant growth in the first 6 months of life. Approximately 5,280 pregnant women will be enrolled into the study from 12 health centers in the Amhara region of Ethiopia. Routine antenatal care will be strengthened in all health centers, and six health centers will be randomized to additionally provide a nutritional intervention including daily multiple-micronutrient or a fortified balanced-energy protein supplement for malnourished women. Women across all 12 health centers will be individually randomized to receive one of three infection management interventions in pregnancy: 1) enhanced infection management package (screening-treatment for urinary tract infections and sexually transmitted infections, presumptive deworming); 2) presumptive azithromycin (2g at <24 wks and a second dose at least 4 weeks later); or 3) placebo. The women and their infants will be followed until 6 months postpartum. Outcomes of interest include birth size (weight, length), gestational age, maternal weight gain in pregnancy, maternal anemia, antimicrobial resistance, and infant size at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women <=24 weeks gestation with a viable pregnancy based on a best clinical algorithm (LMP and/or symphysis fundal height)

Exclusion Criteria:

* Pregnant women presenting at enrollment >24 weeks
* Pregnant women presenting with non-viable fetus
* Women who do not intend to deliver in the study catchment area
* Known allergy to Azithromycin or macrolide antibiotic
* Women who refuse to provide consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-05-28 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Birth weight | Within 72 hours of birth
  Mean infant weight (g) among live born infants measured <72 hour of delivery
Birth length | Within 72 hours of birth
  Mean infant length (cm) among live born infants measured <72 hours of delivery

SECONDARY OUTCOMES:
Gestational age | Birth
  Mean gestational age at delivery
Preterm birth | Birth
  Proportion of pregnancies resulting in spontaneous birth <37 weeks gestation among all births
Small-for-gestational age (SGA) | within 72 hours of birth
  Proportions of newborns born SGA (<10% birthweight for gestational age and sex) among live born infants whose birthweight if measured within 72 hours of delivery.
Low birthweight | within 72 hours of birth
  Proportion of newborns born with weight <2500 g among liveborn infants whose weight is measured within 72 hours of delivery
Length-for-age | Birth, 6 months
  Mean Length-for-age Z scores at birth and 6 months of age among live born infants based on the WHO growth reference standards (WHO 2006)
Weight-for-age | Birth, 6 months
  Mean Weight-for-age Z scores at birth and 6 months of age among live born infants based on the WHO growth reference standards (WHO 2006)
Rate of weight gain in pregnancy | From date of first 2nd trimester antenatal care (ANC) visit until date of last ANC visit before birth, assessed up to 6 months
  Maternal weight gain (kg) per week gestation in the 2nd and 3rd trimester
Maternal anemia | Third trimester antenatal care visit (28-40 weeks gestation)
  Mean hemoglobin concentration
Stillbirth | Birth
  Rate of stillbirths per 1000 births
Prevalence of nasopharyngeal macrolide resistance in mothers-infants | 1 and 6 months post-partum
  Prevalence of nasopharyngeal macrolide resistance among S. pneumoniae isolates in mothers-infants at 1 and 6 months postpartum

IPD SHARING:
Plan to Share IPD: No